CLINICAL TRIAL: NCT02198573
Title: Molecular Assessment of Artemisinin Resistance Markers, K13 Kelch Propeller and Multi-drug Resistant Gene Polymorphism in Eastern and Western Border Areas of Myanmar
Brief Title: Molecular Assessment of Artemisinin Resistance Markers in Eastern and Western Border Areas of Myanmar
Status: Completed | Type: Observational
Sponsor: Myat Htut Nyunt (Other)
Collaborators: Kangwon National University (Other)
Responsible Party: Sponsor-Investigator, Myat Htut Nyunt, Dr. Myat Htut Nyunt, Department of Medical Research, Lower Myanmar
Organization: Department of Medical Research, Lower Myanmar (Other)
Other Study IDs: WHO_3DF_2013_day3
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Day-3 Positive of Parasitaemia; Prevalence of Drug Resistance Gene Mutation
Keywords: malaria; K13; pfmrp1; Myanmar
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — dried blood spot
Oversight: Data Monitoring Committee: Yes

SUMMARY:
* Artemisinin resistance have been documented in Myanmar and Myanmar artemisinin resistance containment measures have been launched since 2009-2010.
* It is important to monitor the spread and magnitude of artemisinin resistant malaria in Myanmar.
* So, day-3 surveillance study have been conducted.
* Recently artemisinin resistant molecular marker, K13 have been identified and it was used as a tool in this study.

ELIGIBILITY:
Inclusion Criteria:

* confirmed uncomplicated falciparum malaria patients.
* age >2 years
* box sex
* given informed consent

Exclusion Criteria:

* severe malaria
* did not give informed consent
* others diseases

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All of the malaria suspected cases were invited to participated in this study from Myanmar-Thailand border and Myanmar-Bangladesh border.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
day-3 parasite positivity | 3 days
  All of the enrolled patients were monitored with appropriate care up to third day and take the samples on day-3.

SECONDARY OUTCOMES:
Prevalence of the drug resistance marker | up to day-3
  By using the dried blood spots, drug resistance markers were detected by molecular method.

CONTACTS AND LOCATIONS:
Overall Officials: Myat P Kyaw, PhD, Study Director — Department of Medical Research, Lower Myanmar
Locations (1):
- Dr. Myat Phone Kyaw, Yangon, Yangon, Burma

REFERENCES:
- [Background] World Health Organization. World Malaria Report 2013. Geneva, Switzerland, 2013.
- [Background] World Health Organization. Global report on antimalarial efficacy and drug resistance: 2000-2010. Geneva, Switzerland: World Health Organization, 2010.
- [Background] Stepniewska K, Ashley E, Lee SJ, Anstey N, Barnes KI, Binh TQ, D'Alessandro U, Day NP, de Vries PJ, Dorsey G, Guthmann JP, Mayxay M, Newton PN, Olliaro P, Osorio L, Price RN, Rowland M, Smithuis F, Taylor WR, Nosten F, White NJ. In vivo parasitological measures of artemisinin susceptibility. J Infect Dis. 2010 Feb 15;201(4):570-9. doi: 10.1086/650301. PMID 20085495
- [Background] Ariey F, Witkowski B, Amaratunga C, Beghain J, Langlois AC, Khim N, Kim S, Duru V, Bouchier C, Ma L, Lim P, Leang R, Duong S, Sreng S, Suon S, Chuor CM, Bout DM, Menard S, Rogers WO, Genton B, Fandeur T, Miotto O, Ringwald P, Le Bras J, Berry A, Barale JC, Fairhurst RM, Benoit-Vical F, Mercereau-Puijalon O, Menard D. A molecular marker of artemisinin-resistant Plasmodium falciparum malaria. Nature. 2014 Jan 2;505(7481):50-5. doi: 10.1038/nature12876. Epub 2013 Dec 18. PMID 24352242
- [Background] Singh B, Bobogare A, Cox-Singh J, Snounou G, Abdullah MS, Rahman HA. A genus- and species-specific nested polymerase chain reaction malaria detection assay for epidemiologic studies. Am J Trop Med Hyg. 1999 Apr;60(4):687-92. doi: 10.4269/ajtmh.1999.60.687. PMID 10348249
- [Result] Kyaw MP, Nyunt MH, Chit K, Aye MM, Aye KH, Aye MM, Lindegardh N, Tarning J, Imwong M, Jacob CG, Rasmussen C, Perin J, Ringwald P, Nyunt MM. Reduced susceptibility of Plasmodium falciparum to artesunate in southern Myanmar. PLoS One. 2013;8(3):e57689. doi: 10.1371/journal.pone.0057689. Epub 2013 Mar 8. PMID 23520478